CLINICAL TRIAL: NCT00075478
Title: A Multi-center Phase III Study Comparing Nonmyeloablative Conditioning With TBI Versus Fludarabine/TBI for HLA-matched Related Hematopoietic Cell Transplantation for Treatment of Hematologic Malignancies
Brief Title: Total-Body Irradiation With or Without Fludarabine Phosphate Followed By Donor Stem Cell Transplant in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1813.00; NCI-2009-01532 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1813.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA078902 (NIH)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission; Aggressive Non-Hodgkin Lymphoma; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Diffuse Large B-Cell Lymphoma; Hematopoietic and Lymphoid Cell Neoplasm; Indolent Non-Hodgkin Lymphoma; Mantle Cell Lymphoma; Myelodysplastic/Myeloproliferative Neoplasm; Plasma Cell Myeloma; Refractory Chronic Lymphocytic Leukemia; Refractory Hodgkin Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Lymphoma, Large B-Cell, Diffuse; Hematologic Neoplasms; Lymphoma, Mantle-Cell; Myelodysplastic-Myeloproliferative Diseases; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Waldenstrom Macroglobulinemia | interventions — Whole-Body Irradiation; fludarabine phosphate; Mycophenolic Acid; Cyclosporine; Cyclosporins; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (chemotherapy, TBI, transplant, GVHD prophylaxis) (Experimental): Patients receive fludarabine phosphate IV on days -4 to -2. Patients then undergo low-dose TBI on day 0. After TBI, patients undergo PBSCT on day 0. Patients receive cyclosporine PO BID on days -3 to 56 in the absence of GVHD. Patients with no evidence of GVHD at day 56 begin a cyclosporine taper and continue the taper until day 180. Patients with evidence of disease progression and no evidence of GVHD prior to day 56 receive tapered doses of cyclosporine for 2 weeks. Patients also receive MMF PO BID on days 0-28 in the absence of GVHD. If treatment for GVHD is required before day 28, MMF is continued until a steroid taper begins.
  Interventions: Procedure: Total-Body Irradiation; Drug: Fludarabine Phosphate; Drug: Mycophenolate Mofetil; Drug: Cyclosporine; Procedure: Peripheral Blood Stem Cell Transplantation
- Arm II (TBI, transplant, GVHD prophylaxis) (Active Comparator): Patients undergo low-dose TBI on day 0. After TBI, patients undergo PBSCT on day 0. Patients receive cyclosporine PO BID on days -3 to 56 in the absence of GVHD. Patients with no evidence of GVHD at day 56 begin a cyclosporine taper and continue the taper until day 180. Patients with evidence of disease progression and no evidence of GVHD prior to day 56 receive tapered doses of cyclosporine for 2 weeks. Patients also receive MMF PO BID on days 0-28 in the absence of GVHD. If treatment for GVHD is required before day 28, MMF is continued until a steroid taper begins.
  Interventions: Procedure: Total-Body Irradiation; Drug: Mycophenolate Mofetil; Drug: Cyclosporine; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Procedure: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; Total Body Irradiation; Whole-Body Irradiation
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; SH T 586
  Arms: Arm I (chemotherapy, TBI, transplant, GVHD prophylaxis)
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Drug: Cyclosporine — Given PO
  Other Names: 27-400; CsA; Neoral; OL 27-400; Sandimmun
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo transplantation
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation

SUMMARY:
This randomized phase III trial is studying total-body irradiation (TBI) and fludarabine phosphate to see how it works compared with TBI alone followed by donor stem cell transplant in treating patients with hematologic cancer. Giving low doses of chemotherapy, such as fludarabine phosphate, and radiation therapy before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after transplant may stop this from happening. It is not yet known whether TBI followed by donor stem cell transplant is more effective with or without fludarabine phosphate in treating hematologic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival at 3 years after conditioning with 200 cGy TBI alone vs. fludarabine (fludarabine phosphate)/200 cGy TBI in heavily pretreated patients with hematologic malignancies at low/moderate risk for graft rejection.

SECONDARY OBJECTIVES:

I. To compare the non-relapse mortality 1-year after conditioning in patients who received TBI alone vs. fludarabine/TBI.

II. To compare the incidences of graft rejection in patients who received TBI alone vs. fludarabine/TBI.

III. To compare the incidences of grades II-IV acute graft-versus-host disease (GVHD) and chronic extensive GVHD.

IV. To compare rates of disease progression and/or relapse-related mortality.

V. To compare the immune reconstitution and the risks of infections.

OUTLINE:

NONMYELOABLATIVE CONDITIONING REGIMEN: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2. Patients then undergo low-dose TBI on day 0.

ARM II: Patients undergo low-dose TBI on day 0.

ALLOGENEIC PERIPHERAL BLOOD STEM CELL TRANSPLANTATION (PBSCT): After TBI, patients undergo PBSCT on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) twice daily (BID) on days -3 to 56 in the absence of GVHD. Patients with no evidence of GVHD at day 56 begin a cyclosporine taper and continue the taper until day 180. Patients with evidence of disease progression and no evidence of GVHD prior to day 56 receive tapered doses of cyclosporine for 2 weeks. Patients also receive mycophenolate mofetil (MMF) PO BID on days 0-28 in the absence of GVHD. If treatment for GVHD is required before day 28, MMF is continued until a steroid taper begins.

Patients are followed up periodically for 1.5 years and then annually for 5 years post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be not eligible for conventional allogeneic hematopoietic cell transplantation (HCT) and must have disease expected to be stable for at least 100 days without chemotherapy
* An autograft immediately prior (less than 6 months) to nonmyeloablative HCT (tandem approach) is not permitted
* Patients with hematologic malignancies treatable with HCT or with a B cell malignancy except those curable with autologous transplant will be included
* Aggressive non-Hodgkin lymphomas (NHLs) and other histologies such as diffuse large B cell NHL: patients are eligible IF they are not eligible for autologous hematopoietic stem cell transplantation (HSCT), not eligible for conventional myeloablative HSCT, or have failed an autologous HSCT
* Low grade NHL with < 6 month duration of complete remission (CR) between courses of conventional therapy
* Mantle cell NHL; may be treated in first CR
* Chronic lymphocytic leukemia (CLL) must have either:

  * Failed to meet National Cancer Institute (NCI) Working Group criteria for complete or partial response after therapy with a regimen containing fludarabine phosphate (FLU) (or another nucleoside analog, e.g. cladribine [2-CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing FLU (or another nucleoside analog)
  * Failed FLU-cyclophosphamide [CY]-rituximab (FCR) combination chemotherapy at any time point
  * Have "17p deletion" cytogenetic abnormality; patients should have received induction chemotherapy but could be transplanted in 1st CR
  * Or patients with a diagnosis of CLL (or small lymphocytic lymphoma) or diagnosis of CLL that progresses to prolymphocytic leukemia (PLL), or T-cell CLL or PLL
* Hodgkin lymphoma (HL): must have received and failed frontline therapy; patients must have failed or were not eligible for autologous transplant
* Multiple myeloma (MM): must have chemosensitive disease after failed autografting (an autografting immediately prior [within 6 months] to nonmyeloablative HCT [tandem approach] is not permitted)
* Acute myeloid leukemia (AML): must have < 5% marrow blasts at the time of transplant and be beyond first CR
* Acute lymphocytic leukemia (ALL): must have < 5% marrow blasts at the time of transplant and be beyond first CR
* Chronic myelogenous leukemia (CML): patients will be accepted in chronic phase (CP) beyond CP1 if they have received previous myelosuppressive chemotherapy or HCT, < 5% marrow blasts at time of transplant
* Myelodysplastic syndromes (MDS)/myeloproliferative disorders (MPD): must have received previous myelosuppressive chemotherapy or HCT, < 5% marrow blasts at time of transplant
* Waldenstroms Macroglobulinemia: must have failed 2 courses of therapy
* Patients will not be allowed to receive myelosuppressive chemotherapy for three weeks prior to conditioning
* Patients < 12 years old must be approved by both the participating institutions' patient review committee such as the Patient Care Conference (PCC) at the Fred Hutchinson Cancer Research Center (FHCRC) and the FHCRC principal investigator
* Patients who refused to be treated on a conventional HCT protocol; for this inclusion criterion, transplants must be approved by both the participating institution's patient review committee such as the Patient Care Conference (PCC) at the FHCRC and the FHCRC principal investigator
* Patients with human leukocyte antigen (HLA)-matched related donors
* DONOR: Related donor who is HLA genotypically identical at least at one haplotype and may be phenotypically or genotypically identical at the allele level at HLA-A, -B, -C, -DRB1, and -DQB1
* DONOR: Donor must consent to filgrastim (G-CSF) administration and leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)
* DONOR: For females of child bearing age, serum pregnancy qualitative (PGSTAT) within 72 hours prior to initial dose of filgrastim (G-CSF); results must be available prior to filgrastim

Exclusion Criteria:

* Eligible for a high priority curative autologous transplant
* Patients with rapidly progressive, aggressive NHL unless in minimal disease state
* Patients with chronic myelomonocytic leukemia
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with AML, ALL or CML
* Life expectancy severely limited by diseases other than malignancy
* Any current central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Fertile men or women unwilling to use contraceptives during and for up to 12 months post treatment
* Female patients who are pregnant or breastfeeding
* Human immunodeficiency virus (HIV) positive patients
* Patients with active non-hematological malignancies (except localized non-melanoma skin malignancies)
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence
* Fungal infections with radiological progression after receipt of amphotericin formulation or mold-active azoles for greater than 1 month
* Patients with active bacterial or fungal infections unresponsive to medical therapy
* Karnofsky score < 50 for adult patients
* Lansky-Play performance score < 50 for pediatric patients
* The addition of cytotoxic agents for "cytoreduction" with the exception of tyrosine kinase inhibitors (imatinib mesylate), cytokine therapy, hydroxyurea, low dose cytarabine, chlorambucil, or rituxan will not be allowed within three weeks of the initiation of conditioning
* Patients with the following organ dysfunction:

  * Symptomatic coronary artery disease or ejection fraction < 35% or other cardiac failure requiring therapy (required for patients with history of cardiac disease or anthracycline use); ejection fraction is required if age > 50 years or there is a history of anthracycline exposure or history of cardiac disease
  * Poorly controlled hypertension on multiple antihypertensives
  * Pulmonary: diffusion capacity of carbon monoxide (DLCO) < 30%, total lung capacity (TLC) < 30%, forced expiratory volume in one second (FEV1) < 30% and/or receiving supplementary continuous oxygen; the FHCRC study principal investigator (PI) must approve enrollment of all patients with pulmonary nodules
  * Liver function abnormalities: patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease
* DONOR: Age less than 12 years
* DONOR: Identical twin
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Known allergy to filgrastim
* DONOR: Current serious systemic illness that would result in increased risk for filgrastim mobilization and harvest of PBSC

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2003-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (10):
- United States (6):
  - OHSU Cancer Institute-Southern Region, Medford, Oregon
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (3):
  - Medizinische Univ Klinik Koln, Cologne
  - Universitaet Leipzig, Leipzig
  - University of Tuebingen-Germany, Tübingen
- University of Torino, Torino, Italy

REFERENCES:
- [Background] Kornblit B, Maloney DG, Storb R, Storek J, Hari P, Vucinic V, Maziarz RT, Chauncey TR, Pulsipher MA, Bruno B, Petersen FB, Bethge WA, Hubel K, Bouvier ME, Fukuda T, Storer BE, Sandmaier BM. Fludarabine and 2-Gy TBI is superior to 2 Gy TBI as conditioning for HLA-matched related hematopoietic cell transplantation: a phase III randomized trial. Biol Blood Marrow Transplant. 2013 Sep;19(9):1340-7. doi: 10.1016/j.bbmt.2013.06.002. Epub 2013 Jun 11. PMID 23769990
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Started | 42 | 45
Completed | 41 | 44
Not Completed | 1 | 1
Not completed — not eligible | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomization will be stratified on institution, disease risk (indolent vs. aggressive), and prior conventional HCT and will be balanced (blocked) over time.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis) | Total
Number analyzed (Participants) | 41 | 44 | 85
Age, Continuous [Median (Full Range); unit: years] | 57 [18 to 72] | 54.5 [18 to 74] | 56 [18 to 74]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 36 | 37 | 73
  >=65 years | 4 | 6 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 25 | 33 | 58
Region of Enrollment [Number; unit: participants]
  United States | 33 | 37 | 70
  Germany | 6 | 6 | 12
  Italy | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Percentage of patients surviving as estimated by Kaplan-Meier.
Time Frame: 3 years after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 41 | 44
percentage of participants | 65 | 54
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) vs Arm II (TBI, Transplant, GVHD Prophylaxis); Reference arm is Arm 2; Test type: Superiority or Other; p = .09, Regression, Cox; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.3 to 1.1]

2. Secondary Outcome: Incidence of Non-relapse Mortality
Description: Percentage of NRM as estimated by cumulative incidence methods with competing risks
Time Frame: 3 years after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 41 | 44
percentage of participants | 7 [9 to 254] | 9 [98 to 287]
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) vs Arm II (TBI, Transplant, GVHD Prophylaxis); Test type: Superiority or Other; p = 0.59, Regression, Cox; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.1 to 3.0]

3. Secondary Outcome: Incidence of Relapse/Progression
Description: Percentage of relapse estimated by cumulative incidence methods
Time Frame: 3 years after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 41 | 44
percentage of participants | 40 | 55
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) vs Arm II (TBI, Transplant, GVHD Prophylaxis); Test type: Superiority or Other; p = 0.06, Regression, Cox; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.3 to 1.0]

4. Secondary Outcome: Incidence of Relapse-related Mortality
Description: Percentage of death following relapse/progression, estimated by cumulative incidence methods
Time Frame: 3 years after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 41 | 44
percentage of participants | 28 | 37
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) vs Arm II (TBI, Transplant, GVHD Prophylaxis); Test type: Superiority or Other; p = 0.09, Regression, Cox; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.3 to 1.1]

5. Secondary Outcome: Incidence of Grades II-IV Acute GVHD
Description: Percentage patients with grades II-IV GHVD, estimated by cumulative incidence methods
Time Frame: 120 days after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 41 | 44
percentage of participants | 46 | 32
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) vs Arm II (TBI, Transplant, GVHD Prophylaxis); Test type: Superiority or Other; p = 0.16, Regression, Cox; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [0.8 to 3.1]

6. Secondary Outcome: Incidence of Chronic Extensive GVHD
Description: Percentage patients with chronic extensive GVHD, estimated by cumulative incidence methods
Time Frame: 3 years after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 41 | 44
percentage of participants | 72 | 48
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) vs Arm II (TBI, Transplant, GVHD Prophylaxis); Test type: Superiority or Other; p = 0.14, Regression, Cox; Hazard Ratio (HR) = 1.52, 95% CI 2-sided [0.9 to 2.7]

7. Secondary Outcome: Incidence of Graft Rejection
Description: Donor CD3 chimerism less than 5%
Time Frame: 1 year after transplant
Measure: Number; unit: participants
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 41 | 44
participants | 0 [0 to 0] | 2 [31 to 31]

8. Secondary Outcome: Progression-free Survival
Description: Percentage of patients with progression-free survival, estimated by cumulative incidence methods
Time Frame: 3 years after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 41 | 44
percentage of participants | 53 | 36
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) vs Arm II (TBI, Transplant, GVHD Prophylaxis); Test type: Superiority or Other; p = 0.05, Regression, Cox; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.3 to 1.0]

ADVERSE EVENTS:
Arm/Group | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) | Arm II (TBI, Transplant, GVHD Prophylaxis)
Serious Adverse Events (participants affected / at risk) | 8/41 | 5/44
Other Adverse Events (participants affected / at risk) | 34/41 | 20/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) (N=41) | Arm II (TBI, Transplant, GVHD Prophylaxis) (N=44)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
seizure (Nervous system disorders) | 1 | 0
pericardial effusion (Cardiac disorders) | 1 | 0
thrombosis (Vascular disorders) | 2 | 1
Bactrim anaphylaxis (Immune system disorders) | 1 | 0
Graft versus host disease with infection and organ failure (Immune system disorders) | 0 | 2
subdural hematoma (Vascular disorders) | 0 | 1
sepsis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemotherapy, TBI, Transplant, GVHD Prophylaxis) (N=41) | Arm II (TBI, Transplant, GVHD Prophylaxis) (N=44)
Blood/Bone marrow (Blood and lymphatic system disorders) | 15 | 10
Cardiovascular (Cardiac disorders) | 4 | 5
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Gastrointestinal (Gastrointestinal disorders) | 2 | 3
Hemorrhage (Vascular disorders) | 3 | 1
Hepatic (Hepatobiliary disorders) | 5 | 3
Metabolic/Laboratory (Metabolism and nutrition disorders) | 3 | 1
Pain (General disorders) | 1 | 0
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Renal/Genitourinary (Renal and urinary disorders) | 4 | 1
Second Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes